CLINICAL TRIAL: NCT07097194
Title: Be A Quitter: Illinois Small Business EX Program Dissemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21520
Record Dates: First submitted 2022-07-18; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EX program participant (Experimental): Individual who signs up for digital tobacco cessation program (EX program)
  Interventions: Behavioral: EX program

INTERVENTIONS:
Behavioral: EX program — Quit plan with interactive exercises, educational videos, and tailored text messages and emails; peer support; coach chatting; nicotine replacement therapy (patches, gum, or lozenges). All components are self-selected.

SUMMARY:
Disseminate the EX tobacco cessation program to Illinois small businesses

DETAILED DESCRIPTION:
This project is designed to provide small businesses throughout Illinois the opportunity to provide a proven tobacco cessation program to their employees at no or reduced cost to the business. The investigators will examine practices that facilitate dissemination of the program, employee usage, as well as benefits of enrollment for individual's mental health, workplace functioning, and family relationships.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Illinois
* 18 years of age or older
* Current tobacco user
* Seeking to quit tobacco use and willing to participate in the EX program
* Willing to answer surveys at 5 occasions over the course of a year
* Employed at collaborating business in Illinois

Exclusion Criteria:

* Not employed at collaborating business in Illinois

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Participant enrollment | Through study completion, an average of 1 year
  Number of individuals that enroll
Quit planning | Through study completion, an average of 1 year
  Number of steps completed for quit plan
Business enrollment | Through study completion, an average of 1 year
  Number of businesses that enroll

SECONDARY OUTCOMES:
General Quality of Life | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  1 item quality of life measure from World Health Organization brief quality of life assessment (1-5, higher is better quality of life)
General Health | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  4 items from RAND (Research and Development) Corporation Short Form Health Survey (1-4, higher is better health)
Work functioning | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  1 item of general ability to function at work (1-5 scale, higher is better working functioning)
Exercise | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  1 item of frequency of exercise (1-6, higher is more weekly exercise)
Psychological distress | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  Kessler 6 item psychological distress (1-5, higher is more distress)
Alcohol Use | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  PROMIS (Patient-Reported Outcomes Measurement Information System) 7 item problematic alcohol use (1-5, higher is more problematic alcohol use)
Anger | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  NIH PROMIS 5 item anger measure (1-5, higher is more anger)
Couple Relationship Satisfaction | Baseline, 3 month, 6 month, 9 month, and 12 month follow-up
  4 item Couple Satisfaction Index (3-21 [summed score], higher is more satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Extension, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No